CLINICAL TRIAL: NCT03972566
Title: Localized Effects of Photobiomodulation and Exogenous Nitric Oxide on CREST Patients Calcinosis Cutis & Raynaud Phenomenon
Brief Title: Localized Effects of PBM and Exogenous NO on CREST Patients Calcinosis Cutis & Raynaud Phenomenon
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RoseLab Skin Optics Laboratory (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Dr Daniel Barolet, Director, RoseLab Skin Optics Laboratory
Other Study IDs: NO-5420
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: CREST Syndrome; Calcinosis Cutis; Raynaud Phenomenon
Keywords: Nitric Oxide; Photobiomodulation; LLLT; Photomedicine
MeSH Terms: conditions — CREST Syndrome; Calcinosis Cutis; Raynaud Disease | interventions — Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Gaseous NO emanating from subject's arms, Digital Thermal Monitoring (DTM) to measure vascular reactivity
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CREST with Calcinosis cutis
  Interventions: Drug: INOMAX
- CREST without Calcinosis cutis
  Interventions: Drug: INOMAX

INTERVENTIONS:
Drug: INOMAX — INOMAX + PBM

SUMMARY:
Background CREST is an acronym for the cardinal clinical features of the syndrome (Calcinosis, Raynaud phenomenon, Esophageal dysmotility, Sclerodactyly, and Telangiectasia) and part of the heterogeneous group of sclerodermas.

Calcinosis is the pathologic calcification of soft tissues. When symptomatic, they can be tender and painful, ulcerate, and drain a white chalky substance. With time, heterotopic bone formation may occur. Inflammatory reactions also intermittently occur at the site of calcinosis. It has been suggested that TGF-beta3 plays a major role in the pathogenesis of calcinosis.

A variety of medical therapies have been used to try to alleviate patient symptoms. These include pharmacological approaches (e..g., warfarin), surgical curettage or excision, as well as carbon dioxide laser treatments. No consistently reliable pharmacological treatment seems to be available to prevent or eliminate calcinosis. Curettage and excision and carbon dioxide laser of localized painful large deposits can relieve symptoms but recurrence is common. In addition, aggressive curettage or excision can damage deeper neurovascular structures. While calcinosis is associated with significant morbidity its treatment remains a challenge.

Photobiomodulation (PBM) has been shown to promote wound healing, suppress inflammatory reactions and regulate collagen synthesis in a number of in vitro and in vivo studies.

Human skin contains photolabile nitric oxide (NO) derivatives which decompose after UVA irradiation and release vasoactive NO. However, aside from blue light, barely nothing has been reported about the effects of red and NIR wavelengths.

Method A custom-built air tight sleeve which envelopes the forearm of a subject will be used to measure the NO emanating from the skin under photobiomodulation conditions (red & NIR) and quantified by chemiluminescence detection.

Simultaneously, CREST patient's hands exhibiting calcinosis and/or Raynaud phenomenon will be exposed to exogenous gaseous nitric oxide (INOMAX) to determine the vascular impact of this approach.

This case series will assess Light Emitting Diode (LED) based PBM therapy as a treatment alternative for cutaneous calcinosis and the effects of gaseous NO on calcinosis and/or Raynaud phenomenon in CREST patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-60 years of age
* CREST syndrome with calcinosis cutis.
* CREST syndrome without calcinosis cutis.

Exclusion Criteria:

* Diabetes mellitus
* Acute inflammation
* Arrhythmia
* Acute malignancy
* Renal failure
* Active CVD
* Photodermatosis and/or photosensitivity including skin cancer-prone disease/syndrome (XP and Bloom Syndrome)
* Porphyria and/or hypersensitivity to porphyrins
* Congenital or acquired immunodeficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering from CREST that have consulted in Dr. Barolet's Clinic of Dermatology
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2019-06-20 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Chemiluminescence detection | 15 minutes
  Sievers Nitric Oxide Analyzer NOA 280i detects [NO] in Ambient Air or Solution
Endothelial Measurement | 5 minutes
  VENDYS II

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Dr Daniel Barolet, Laval, Quebec, Canada